CLINICAL TRIAL: NCT02385734
Title: Concentrated Growth Factor Membrane in the Treatment of Adjacent Multiple Gingival Recessions: A Split Mouth Randomized Clinical Study
Brief Title: Concentrated Growth Factor in the Treatment of Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Seyma Bozkurt Doğan, Şeyma Bozkurt Doğan, Asisstant Proffessor, Bulent Ecevit University,, Bulent Ecevit University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-62550515-03
Record Dates: First submitted 2015-03-02; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Gingival Recession
Keywords: Multiple gingival recession; Concentrated growth factor; Coronally advanced flap
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Concentrated growth Factor Membrane (Experimental): Autogenous platelet and leukocyte fibrin material was obtained from blood.
  Interventions: Other: Concentrated Growth Factor Membrane; Procedure: Coronally Advanced Flap
- Coronally Advanced Flap (Active Comparator): Periodontal plastic surgery procedure in the treatment of gingival recession
  Interventions: Procedure: Coronally Advanced Flap

INTERVENTIONS:
Other: Concentrated Growth Factor Membrane — Concentrated growth factor membrane is produced by the centrifugation of venous blood and platelets are concentrated in a gel layer containing fibrin matrix
  Other Names: An agent of platelet concentrates
  Arms: Concentrated growth Factor Membrane
Procedure: Coronally Advanced Flap — Periodontal plastic surgery technique

SUMMARY:
This study hypothesized that Concentrated Growth Factors'(CGF) placement together with Coronally Advanced Flap (CAF) may enhance the healing of soft tissues. Therefore, the aim of this study was to determine the clinical effect of CGF combination with CAF compared to CAF alone in the treatment of adjacent multiple gingival recessions.

DETAILED DESCRIPTION:
The gingival recessions have been successfully treated by several periodontal plastic surgery procedures. Among the different types of procedures used, Coronally Advanced Flap (CAF) was the most frequent approach, and when combined with a connective tissue graft is accepted as a gold standard therapy. Recently, investigators reported the use of CGF in the reconstruction of bone defects. They concluded that bone formation had significantly increased by using CGF It has been used to accelerate new bone formation associated with guided bone regeneration in sinus augmentation.They stated that CGF may have a better regenerative capacity and high versatility. Therefore, this study hypothesized that CGFs' placement together with CAF may enhance the healing of soft tissues. Therefore, the aim of this study was to determine the clinical effect of CGF combination with CAF compared to CAF alone in the treatment of adjacent multiple gingival recessions.

The patients of this randomized, split mouth and controlled clinical trial study protocol were selected from individuals referred to the Department of Periodontology, at Faculty of Dentistry, Bülent Ecevit University, for either dentin hypersensitivity or aesthetic complaints between April 2013 and April 2014.

All the subjects received oral hygiene instructions and full-mouth scaling were performed 1 month before surgery. They were instructed to perform a non-traumatic brushing technique (Roll) using an ultra soft toothbrush. In twenty subjects (mean age 37.10 ±1.03, 20-45years, 13 females, 7 males), one side of the jaw received CAF (control sites)( 59 defects), the opposite site received CAF+CGF (test sites) (60 defects).

Full-mouth Plaque index and Gingival index were evaluated before surgery. Custom acrylic guides were fabricated to measure the clinical parameters at the mid-buccal aspect of the treated teeth.Probing depth (PD), Clinical Attachment Loss (CAL),Recession Depth (RD),Keratinized Gingiva Width (KGW) were recorded at the mid-buccal aspect of the treated teeth. Gingival Thickness (GT) was evaluated mid-facially, 2mm apical to the gingival margin at the attached gingiva or the alveolar mucosa, using a 20 endodontic reamer attached to a rubber stopper under the local anesthesia. After carefully removing the reamer, GT was measured with a digital caliper with 0.05 resolution PD, CAL, RD, KGW and GT were assessed at baseline and 6th months. Complete root coverage (CRC)and Percentage Root Coverage(PRC) were calculated at 6th months.

Intravenous blood was collected and placed into two different a 10mL glass-coated plastic tube without anticoagulant solutions. These tubes were then immediately centrifuged with a CGF centrifuge machine. The CGF clot was removed from the tube and separated from the Red Blood Cell by using microsurgical scissors. The CGF was squeezed in a special box that produces membranes at a constant thickness of 1mm.CGF membrane was immediately placed over the recession area.

All surgeries were performed by the same expert periodontist during a single surgical session Gingival recession sites were randomly determined as either test or control site by tossing a coin immediately before the surgical procedure.

Sutures were removed after 10 days and plaque control was maintained by CHX for additional 2 weeks. The patients started brush the tooth at the end of the 3rd week and they were again instructed in mechanical tooth cleaning of the treated tooth using an ultra soft toothbrush and roll technique. Oral hygiene instructions were provided at each postoperative visit.

ELIGIBILITY:
Inclusion Criteria:

* systemically and periodontally healthy,
* non-smokers
* presence of ≥ 2 buccal adjacent Miller Class I and II gingival recession with ≥ 2 mm gingival recession depth , probing depth <3 mm and gingival thickness (GT) ≥ 1 mm on both sides of the maxillary arch
* width of keratinized gingiva ≥ 2mm
* presence of identifiable cemento-enamel junction
* full-mouth plaque index (PI) < 20 % and gingival index (GI) scores <1,
* presence of tooth vitality and absence of caries, restorations and furcation involvement in the treated area,

Exclusion Criteria:

* patients who had systemic problems that wound contraindicate for periodontal surgery, - usage of medications known to interfere with healing and to cause gingival enlargement - recession defects associated with demineralization, deep abrasion,
* previous surgery in the defects area within the past 1 year,
* pregnant or lactating females
* drug and alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Complete root coverage | 6 months
  Change from baseline in percentage of complete root coverage at 6th months.

SECONDARY OUTCOMES:
Percentage root coverage | 6 months
  Change from baseline in percentage of root coverage at at 6th months.
Keratinized gingiva width | 6 months
  The distance is from the mucogingival junction (MGJ) to the gingival margin
Recession depth | 6 th months
  The distance is from the cemento-enamel junction to the gingival margin
Gingival Thickness | 6 months
Probing depth | 6 months
  The distance is from the gingival margin to the bottom of the sulcus
Clinical attachment loss | 6 months
  The distance is from the cemento-enamel junction to the bottom of the sulcus.